CLINICAL TRIAL: NCT04787133
Title: Assessment of the Perioperative Experience of Patients According to Different Preoperative Anesthesia Consultation (PAC) Modalities
Brief Title: Supervised Nurse Assisted Preoperative Assessment (SNAP)
Acronym: SNAP
Status: Withdrawn | Type: Observational
Why Stopped: budgetary reason
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: JDS_2020_29
Record Dates: First submitted 2021-01-26; First posted 2021-03-08 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Satisfaction, Patient; Surgery
Keywords: Anesthesia consultation; Patient satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Compare the experience of patients receiving an "optimized" preoperative anesthesia consultation (PAC) performed by a Nurse Anesthetist (supervised by an anesthetist) to those receiving a "standard" CSA ( CSA by an anesthetist alone).

DETAILED DESCRIPTION:
Preoperative anesthesia consultations (PACs) are a key moment in the perioperative care journey. During the PAC, the doctor assesses the patient's state of health (allowing an assessment of the perioperative risk), establishes the anesthesia protocol and writes the preoperative prescriptions. PAC also helps inform and educate patients to reduce their anxiety.

Indeed, if the perioperative care pathway and the risks associated with anesthesia are poorly understood, there is an increased risk of preoperative anxiety, poor compliance with preoperative prescriptions, and therefore potential cancellation of the surgical intervention.

In many countries, preoperative PACs are performed by nurses trained and supervised by anesthetists. These PACs take longer than a consultation carried out by a doctor alone, but would on the one hand have a positive effect on patient education and, on the other hand, ultimately reduce the time and costs associated with the PAC . On the other hand, the impact of PACs performed by nurses supervised by physicians on the perioperative experience of patients and on the rate of cancellations of scheduled interventions has not yet been demonstrated.

Since 2013, so-called "optimized" consultations (PAC carried out by a state-certified nurse - IDE - supervised by an anesthesiologist) have been carried out at the Adolphe de Rothschild Foundation (Paris), for patients having a scheduled surgery intervention. cataract under locoregional or general anesthesia. First, the IDE collects the patient's history and treatments and informs him of the perioperative care pathway. In a second step, the doctor performs the pre-anesthetic medical examination, completes the medical examination and writes the appropriate pre and postoperative prescriptions. This method of consultation made it possible to optimize medical time while providing complete, even better, information to the patient.

That is why optimized PACs may improve the patient's perioperative experience and reduce preoperative cancellations regardless of the type of surgery. programmed.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old
* Must benefit from an anesthesia consultation for general or regional anesthesia for scheduled surgery, whatever it is.
* Express consent to participate in the study
* Affiliate or beneficiary of a social security scheme

Exclusion Criteria:

* Patient benefiting from a legal protection measure
* Pregnant or breastfeeding woman
* Patient unable to understand and read French, as well as to complete a self-administered questionnaire
* Patient with mental retardation with impaired judgment

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients who will have an anesthesia consultation on one of the randomized shifts
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-02 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Assessment of patient satisfaction with a perioperative anesthetic evaluation | 48 hours
  Patient satisfaction will be assess within 48h after surgery using the "Evaluation du Vécu de l'Anesthésie" or "EVAN" (EVAN-G for EVAN-General anesthesia or EVAN-LR for EVAN-locoregional anesthesia).
  The EVAN-G includes 26 items; six specific scores (Attention, Information, Discomfort, Privacy, Waiting and Pain) and one global index score. The EVAN-LR comprises 19 items; ﬁve specific scores (Attention, Information, Discomfort, Waiting, and Pain) and one global index score.
  Specific and global index scores were linearly transformed to a 0-100 scale, with 100 indicating the best possible level of satisfaction and 0 indicating the worst.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Fondation Adolphe de Rothschild, Paris, Île-de-France Region, France